CLINICAL TRIAL: NCT01991899
Title: Study of Immunogenicity, Reactogenicity and Safety of the Combined Measles, Mumps and Rubella Vaccine Produced by Bio-Manguinhos/Fiocruz in Children 12-15 Months of Age, Followed by Tetraviral Vaccine in Children 15-18 Months.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz) (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: ASCLIN/002/2013
Record Dates: First submitted 2013-11-08; First posted 2013-11-25 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Measles; Mumps; Rubella; Varicella
Keywords: Measles, mumps and rubella vaccine; Tetraviral vaccine; Immunogenicity, Reactogenicity and Safety; Consistency of production
MeSH Terms: conditions — Measles; Mumps; Rubella; Chickenpox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MMR Bio-Manguinhos (Experimental): Arm 1:1170 children will receive MMR Bio-Manguinhos, 3 diferents lots
  Interventions: Biological: MMR Bio-Manguinhos
- MMR GlaxoSmithKline (Active Comparator): Arm 2:390 children will receive MMR GlaxoSmithKline
  Interventions: Biological: MMR GlaxoSmithKline

INTERVENTIONS:
Biological: MMR Bio-Manguinhos — 1170 children will receive 100% produced by Bio-Manguinhos, 3 diferents lots. Application of a 0.5 ml dose, subcutaneous 390 children will receive 0,5 ml, subcutaneous, MMR GlaxoSmithKline
  Other Names: MMR GlaxoSmithKline
  Arms: MMR Bio-Manguinhos
Biological: MMR GlaxoSmithKline — 390 children will receive 0,5 ml MMR GlaxoSmithKline
  Other Names: MMR Bio-Manguinhos
  Arms: MMR GlaxoSmithKline

SUMMARY:
It is a clinicaltrial Phase III , randomized, double -blind , 4-arm (390 each one):

This study will include 1560 children and will use 3 batches of vaccine produced by Bio - Manguinhos with viral bulk of GSK combined measles , mumps and rubella applied in healthy children 12-15 months of age, and 01 batch of MMR to reference( GSK ), applied in healthy children aged 12-15 months old . The vaccine is administered as MMR 1st dose.

Two hypotheses are tested :

1. Consistency of production ( equivalence between batches )of 3 batches of vacines(TV1, TV2 , TV3 Bio- Manguinhos). Noninferiority vaccine Bio TV (Fiocruz, Rio de Janeiro), ie, the measles, mumps and rubella in Brazil is as immunogenic and safe as the measles, mumps and rubella reference, already used in routine NIP (production Bio-Manguinhos/FIOCRUZ with viral concentrate, bulk, GSK).

   The MMR vaccine (Bio-TV) will have the same composition (vaccine strains) and the same method of production of MMR (TV-GSK): Wistar RA27 / 3 rubella, Schwarz strain of measles vaccine, and strain RIT 4385 - derived from the Jeryl Lynn strain of mumps vaccine.

   As 2nd dose, children receive the vaccine tetraviral measles-mumps-rubella-varicella, aged 15-18 months, according to the guidance of the National Immunization Program.
2. Noninferiority vaccine Bio TV (Fiocruz, Rio de Janeiro):the measles, mumps and rubella vaccine in Brazil is as immunogenic and safe as the measles, mumps and rubella reference, already used in routine NIP (production Bio-Manguinhos/FIOCRUZ with viral concentrate, bulk, GSK).

Returns for blood sampling will be scheduled for 51 days, ranging from 42 to 60 days after dose of MMR vaccine dose and after tetraviral. We will colect the firt blood sample before the first vaccination too.

It will describe the major adverse events observed after vaccination , comparing their frequency in groups of MMR vaccine with the Brazilian reference vaccine .

DETAILED DESCRIPTION:
Status:Not yet recruiting: participants are not yet being recruited

Parents or guardians, potential participants to the study, will be identified by the field staff of the project and invited to an interview host, which will be presented in the study objectives, the necessary procedures (vaccine, blood collection and pre-vaccination postvaccination, interviews, etc..), their frequency, duration, benefits and risks of the study. It will also read and discussed the Informed Consent Form (ICF).

It will be made Serology, pre-and post-vaccination, using the technique of enzyme immunoassay (ELISA DadeBehring / SIEMENS) for measles, rubella, mumps and varicella, with titration of specific IgG antibodies in the Laboratory of Respiratory Virus / IOC / Fiocruz;

Titration of neutralizing antibodies to measles and mumps, pre and post vaccination (by Plaque Reduction Neutralization Test, PRNT) in samples that are successful seronegative. Will be held at LATEV / Bio-Manguinhos / Fiocruz.

Control of adverse events after application of vaccine will be made by means of annotations that should be completed by a responsible journal and analyzed by the doctor. They will be have a number phone 24 hours to contact with the doctor.

The monitors will visit the initiation of the study (day 0), regular visits during the study and a visit closing soon after completion of the study. Monitors should review the FRC, comparing them with source documents to verify the accuracy of data collection, assess adherence to good clinical practice and ensure that the study data are complete, accurate and integers. Monitors should make sure of the existence of time, space and qualified personnel in the days of monitoring visits.

Plan for data analysis

The consistency of production batches (equivalence) .Upper and lower limits of the confidence intervals of 95% of the difference in seroprotection results for each of the three pairs of contrasting antigens lots (three batches compared in pairs) between -10% and +10%, two-tailed analysis.

. ratio of the geometric mean titers for each of the antigens between 0.5 and 2. The 3 lots will be considered to be consistent in terms of TMG to a particular vaccine component, if all three 95% CI of the ratio of two-tailed paired TMG are between 0.5 and 2.

Non-inferiority

* Difference seroprotection for each of the antigens in the vaccines under test and reference vaccines or greater - 10%, one-tailed analysis. More precisely, the lower limit of 95% of the difference between the seroprotection rates in the vaccine test and reference vaccine should be greater than 10% (e.g. 4%, -3%, etc. .)
* ratio of the geometric mean titers for each of the antigens ≥ 0.5 (for vaccines and vaccine Bio-Manguinhos reference).

The analysis of non-inferiority will take into account three batches of vaccines TV1, TV2, TV3 and that will be compared together with the reference vaccine, if any consistency of production batches.

This procedure is performed in the 2nd serology after vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Children of both sexes
* Age between 12 to 15 months .
* Child in good health , without significant past medical history personal , such as genetic syndromes , epilepsy , diabetes , severe infections and immune dysfunctions .
* Consent of father or mother , or legal guardian of the child to participate in the study and signing the Informed Consent Form.
* Disposition of the father or mother, or legal guardian to provide name, address, phone and other information so you can get in touch with this, if necessary .
* The responsible person be able to understand the risks of the experimente
* The responsible person be able to understand and sign the informed consent form . If the charge is not able to sign ( illiterate ) the IC may be signed by an impartial witness who has followed the entire procedure .
* Availability return to collect post-vaccination - The research subjects may not be participating in another clinical study during this study.
* Not having received injectable live virus vaccine in the last 30 days.

Exclusion Criteria:

* - Children with a history of measles, rubella and / or mumps .
* Have received MMR or tetraviral previously documented in book vaccination ( eg . : In situations of conducting national campaign or blocking vaccination before suspected cases ).
* Have received a blood transfusion , including immunoglobulins , less than 1year .
* Skin lesions at sites of venipuncture .
* Child subject to abnormal bleeding after injections .
* Using the last 6 months at doses of corticosteroids and other immunosuppressive immunosuppressants.
* Fever on the day of inclusion or in the 3 days prior to the inclusion in this case may be rescheduled for inclusion 14 days after fever subsides .
* Antibiotic use on the day of inclusion or in the last 7 days prior to inclusion - in this case , may be rescheduled for inclusion after 14 days from the last day of antibiotic use .
* Significant abnormality on physical examination the day of enrollment . Known systemic hypersensitivity to neomycin or any other component of the vaccine .
* Individuals with a history of severe allergy , anaphylaxis to egg proteins .
* Have received live attenuated vaccine , as the vaccine for yellow fever in the 30 days prior to vaccination with MMR and the 2nd and 3rd collections .

Ages: 12 Months to 18 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1560 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Immunogenicity comparing the 3 lots of MMR vaccine produced totally in Brazil and reference vaccine. | Thirty days after MMR vaccine
  Difference seroprotection for each of the antigens in the vaccines under test and reference vaccines or greater - 10%, one-tailed analysis. More precisely, the lower limit of 95% of the difference between the seroprotection rates in the vaccine test and reference vaccine should be greater than 10% (e.g. 4%, -3%, etc. .) evaluate the immunogenicity• Ratio of the geometric mean titers for each of the antigens ≥ 0.5 (for Bio-Manguinhos vaccine and reference vaccine).
  The analysis of non-inferiority will take into account three batches of vaccines TV1, TV2, TV3 and that will be compared together with the reference vaccine, if any consistency of production batches.
  This procedure is performed in the 2nd serology after vaccination.
Safety | Thirty days after MMR vaccine
  Parents or guardians will take home the diary for recording adverse events. They will receive training on how to complete the diary of adverse events in health facilities where children are vaccinated after the first dose of MMR. They will receive a ruler and a mercury thermometer to check for adverse events and a pen for note. The diary of adverse events should be completed during the 10 days after vaccination •Adverse events will be compared for each of vaccines (TV1, TV2, TV3 and reference vaccine) and for each dose. Will determine the percentage of subjects with a report of any symptoms (solicited or unsolicited) during the 30 days of follow-up after vaccination. Are tabulated the percentages of subjects with adverse events (for the overall incidence of any symptom, for the incidence of any local symptoms and the incidence of any general symptoms). The comparison between groups will be made by the chi-square test with a significance level of 0.05.
Determine the consistency of production | Thirty days after MMR vaccine
  Difference seroprotection for each of the antigens in the vaccines under test and reference vaccines or greater - 10%, one-tailed analysis. More precisely, the lower limit of 95% of the difference between the seroprotection rates in the vaccine test and reference vaccine should be greater than 10% (e.g. 4%, -3%, etc. .) evaluate the immunogenicity• Ratio of the geometric mean titers for each of the antigens ≥ 0.5 (for Bio-Manguinhos vaccine and reference vaccine).
  The analysis of non-inferiority will take into account three batches of vaccines TV1, TV2, TV3 and that will be compared together with the reference vaccine, if any consistency of production batches.
  This procedure is performed in the 2nd serology after vaccination.

SECONDARY OUTCOMES:
Adverse events after tetraviral | Three months after MMR vaccine
  Describe the major adverse events observed after vaccination.Their parents or guardians will take home the diary for recording adverse events.They will receive a ruler and a mercury thermometer to check for adverse events and a pen for note. The diary of adverse events should be completed during the 10 days after vaccination •Adverse events will be compared for each of vaccines (TV1, TV2, TV3 and reference vaccine) and for each dose. Will determine the percentage of subjects with a report of any symptoms (solicited or unsolicited) during the 30 days of follow-up after vaccination. Are tabulated the percentages of subjects with adverse events (for the overall incidence of any symptom, for the incidence of any local symptoms and the incidence of any general symptoms). The comparison between groups will be made by the chi-square test with a significance level of 0.05.requency in the vaccine groups tetraviral.
Seroconversion after vaccine tetraviral( measles, mumps,rubella and varicela) | Four months after MMM vaccine
  Compare tetraviral seroconversion after MMR vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Eliane Matos Santos, Principal Investigator — The Immunobiological Technology Institute (Bio-Manguinhos) / Oswaldo Cruz Foundation (Fiocruz)
Locations (1):
- Instituto Evandro Chagas, Belém, Pará, Brazil